CLINICAL TRIAL: NCT02371577
Title: A Phase 2 Clinical Trial To Evaluate The Immune Restoration Potential Of Lenalidomide For Patients With CLL-Associated Immunodeficiency
Brief Title: Evaluation of the Immune Restoration Potential Of Lenalidomide
Acronym: Revlimid
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn
Sponsor: University of California, San Diego (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Michael Choi, Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 141671
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Revlimid
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide is administered orally once daily on Days 8-28 of each 28 day cycle. The typical starting dose is 2.5mg PO daily. At the start of each cycle, there is intra-patient dose-escalation to a maximum of 25mg daily, in the absence of grade 2 or higher adverse events.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is administered orally once daily on Days 8-28 of each 28 day cycle. The typical starting dose is 2.5mg PO daily. At the start of each cycle, there is intra-patient dose-escalation to a maximum of 25mg daily, in the absence of grade 2 or higher adverse events Duration of lenalidomide on the clinical trial is for up to 6 cycles, each of 28 day duration.
  Other Names: Revlimid

SUMMARY:
This is phase 2 study of the immunomodulatory drug, lenalidomide, to evaluate potential beneficial effects on the immune system of patients with chronic lymphocytic leukemia (CLL) and CLL-associated immunodeficiency. 17 patients will be enrolled with CLL, small lymphocytic lymphoma (SLL), or monoclonal B-cell lymphocytosis (MBL), and measurable immune compromise, but not an iwCLL indication for CLL therapy (ie non-progressive disease).

DETAILED DESCRIPTION:
This is phase 2 study of the immunomodulatory drug, lenalidomide, to evaluate potential beneficial effects on the immune system of patients with chronic lymphocytic leukemia (CLL) and CLL-associated immunodeficiency. 17 patients will be enrolled with CLL, small lymphocytic lymphoma (SLL), or monoclonal B-cell lymphocytosis (MBL), and measurable immune compromise, but not an iwCLL indication for CLL therapy (ie non-progressive disease). Lenalidomide will be administered orally for 21 days of each 28 day cycle, starting at a 2.5mg dose, with dose escalation each cycle to a maximum of 25mg in the absence of any grade 2 or higher hematologic or non-hematologic adverse events. Treatment duration to primary endpoint assessment is 6 cycles, though patients will not be restricted from continuing lenalidomide off-study, if clinically indicated

ELIGIBILITY:
Main Inclusion Criteria:

1. Clinical and phenotypic verification of B cell CLL/ SLL/ or MBL and measurable disease.
2. Subjects must have total serum IgG < 500 mg/dL
3. Disease Status/ Prior Therapy: There is not any requirement nor restriction for prior therapy.
4. Recovered from the toxic effects of prior therapy to their clinical baseline.
5. Both men and women of all races and ethnic groups are eligible for this trial.
6. Women of childbearing potential (not postmenopausal for at least one year or not surgically incapable of bearing children) must agree not to become pregnant for the duration of the study. Both men and women must agree to use a barrier method of contraception for the duration of the study and until 8 weeks after the final dose of lenalidomide.
7. ECOG performance status of 0-2.
8. Adequate hematologic function:

   8.1. Platelet count ≥ 50,000/µL; AND 8.2. Hemoglobin ≥ 8.0 g/dL 8.3. Absolute neutrophil count > 1000 /uL
9. Adequate renal function:

   9.1. Serum creatinine <1.5 times upper limit of normal; OR 9.2. Calculated Creatinine clearance (CrCl) ≥ 50 mL/min
10. Adequate hepatic function:

    12.1. Total bilirubin ≤ 2.5 times upper limit of normal; AND 12.2. ALT ≤ 2.5 times upper limit of normal.
11. Able to take aspirin (81mg or 325mg) daily, warfarin, low molecular weight heparin, or equivalent anticoagulation as prophylactic medication.
12. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of REMS®.
13. Females of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting Revlimid® and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Revlimid®. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
14. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.

Exclusion Criteria:

1. Progressive CLL requiring therapy based on 2008 international working group guidelines (iwCLL 2008, Hallek et al, Blood 2008).
2. Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
3. Known hypersensitivity to thalidomide or lenalidomide.
4. Prior lenalidomide-associated deep vein thrombosis
5. Deep vein thrombosis or superficial thrombophlebitis of any cause on current anticoagulation therapy at the time of screening.
6. Patients who are currently receiving another investigational agent are excluded.
7. Patients who have had chemotherapy (e.g., purine analogues, alkylating agents), radiation therapy, tyrosine kinase inhibitor therapy, or participation in any investigational drug treatment within 4 weeks of initiation of lenalidomide or at any time during the study.
8. Patients who have had prior (within 8 weeks of initiation of lenalidomide) or concurrent antibody therapy directed against CLL.
9. Current infection requiring parenteral antibiotics.
10. Known seropositive for or active viral infection with human immunodeficiency virus (HIV); or known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) based on detectable viral load. Patients who are seropositive because of hepatitis B virus vaccine are eligible.
11. Active malignancy within the previous 2 years (other than completely resected non-melanoma skin cancer or carcinoma in situ).
12. Known history of IgA or IgG monoclonal gammopathy of undetermined significance (MGUS)
13. Known central nervous system (CNS) involvement by malignancy.
14. Untreated autoimmunity such as autoimmune hemolytic anemia, or immune thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Immunoglobulin G level | 2 years
  IgG levels during and at the completion of 6 months of lenalidomide

SECONDARY OUTCOMES:
Treatment-emergent adverse events, including infections | 2 years
Progression free survival rate at 6 months, determined by International Working Group in CLL (iwCLL) criteria. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — UC San Diego Moores Cancer Center
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States